CLINICAL TRIAL: NCT00000767
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind Trial to Evaluate the Safety and Immunogenicity of a Recombinant Vaccinia-HIV-1 IIIB Env/Gag/Pol Vaccine (TBC-3B)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 014A; 10561 (Registry Identifier: DAIDS ES Registry Number); AVEG 014A/B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Vaccinia Virus; Viral Vaccines; Smallpox Vaccine; HIV-1; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Vaccinia | interventions — Smallpox Vaccine

INTERVENTIONS:
Biological: TBC-3B Vaccine
Biological: Smallpox Vaccine

SUMMARY:
To evaluate, in healthy HIV-1 seronegative vaccinia-immune and vaccinia-naive volunteers, the safety and immunogenicity of an HIV-1 candidate vaccine (TBC-3B) consisting of a live recombinant vaccinia virus expressing the env, gag, and pol genes of HIV-1 IIIB strain. To evaluate the potential of boosting with one of a variety of HIV-1 recombinant subunit, peptide, or pseudovirion vaccines, if available, to augment the immune responses of the vaccinees.

Antigenic drift, defined as the genetic variation of the HIV-1 envelope gene that results in antigenic variation during natural infection, may confound attempts to achieve protective immunity using a vaccine based solely on HIV-1 envelope proteins. Inclusion of conserved core and polymerase proteins along with envelope protein in a candidate vaccine may address some of the problems with antigenic variability. A prime-boost immunization approach using a novel priming immunogen expressing env, gag, and pol genes of the HIV-1 IIIB strain will be attempted in this study.

DETAILED DESCRIPTION:
Antigenic drift, defined as the genetic variation of the HIV-1 envelope gene that results in antigenic variation during natural infection, may confound attempts to achieve protective immunity using a vaccine based solely on HIV-1 envelope proteins. Inclusion of conserved core and polymerase proteins along with envelope protein in a candidate vaccine may address some of the problems with antigenic variability. A prime-boost immunization approach using a novel priming immunogen expressing env, gag, and pol genes of the HIV-1 IIIB strain will be attempted in this study.

In Part I, vaccinia-immune volunteers are randomized to one of two regimens. Group A receives priming with TBC-3B on days 0 and 56, followed by boosting on day 224 (8 months) with one of the following: TBC-3B, an alternative immunogen such as pseudovirion particles or a recombinant HIV-1 subunit or peptide vaccine, or placebo. Group B receives priming with control vaccine (DryVax), followed by boosting with an appropriate placebo. At least 50 percent of subjects in Part I will be observed for a minimum of 8 weeks before subsequent volunteers are enrolled in Part II. PER 11/18/94 AMENDMENT, Part I boosting is given on day 392. PER 5/19/95 AMENDMENT, Part I boosting is given on day 756 if not available on day 392; if the appropriate product is not available then, the study will end on day 756. In Part II, vaccinia-naive volunteers are randomized to one of three regimens. Group C receives TBC-3B on day 0 and saline placebo on day 56. Group D receives TBC-3B on days 0 and 56. Both Group C and D receive boosting with TBC-3B or an alternative immunogen on day 224. Group E receives control vaccine (DryVax) on days 0 and 56, followed by appropriate placebo on day 224. Per 06/10/94 addendum, volunteers will be contacted once or twice per year for at least 5 years to check on health status.

NOTE: Part I (Part A) of the protocol has closed to accrual.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Negative ELISA and Western blot for HIV-1 within 6 weeks prior to immunization.
* Normal history and physical exam.
* History of smallpox vaccination at least 5 years prior to study entry (Part I) OR no prior smallpox vaccination (Part II).
* Absolute CD4 count >= 400 cells/mm3.
* Normal urinalysis.

NOTE:

* No more than 10 percent of volunteers in both Parts I and II may be over 50 years of age.

Exclusion Criteria

Co-existing Condition:

Subjects with the following symptoms or conditions are excluded:

* Positive hepatitis B surface antigen.
* Medical or psychiatric condition (such as recent suicidal ideation or present psychosis) that precludes compliance.
* Occupational responsibilities that preclude compliance.
* Active syphilis. NOTE: Subjects with serology documented to be a false positive or due to a remote (> 6 months) treated infection are eligible.
* Active tuberculosis. NOTE: Subjects with a positive PPD and a normal chest x-ray showing no evidence of TB and not requiring isoniazid therapy are eligible.
* Eczema.
* Household contact with persons meeting any of the following criteria:
* pregnancy, less than 12 months of age, eczema, immunodeficiency disease, or use of immunosuppressive medications.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, autoimmune disease, or use of immunosuppressive medications.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* Eczema within the past year.
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g., Steven-Johnson syndrome, bronchospasm, or hypotension).
* Prior psychiatric condition (such as history of suicide attempts or past psychosis) that precludes compliance.
* History of cancer unless there has been surgical excision that is considered to have achieved cure.

Prior Medication:

Excluded:

* Prior HIV vaccines.
* Live attenuated vaccines within the past 60 days. NOTE: Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) do not exclude but should be administered at least 2 weeks prior to HIV immunizations.
* Experimental agents within the past 30 days.

Prior Treatment:

Excluded:

* Receipt of blood products or immunoglobulins within the past 6 months. It is STRONGLY RECOMMENDED that any activity that might expose subject to HIV (unprotected sex or needle sharing) be avoided.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Study Completion 1996-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keefer M, Study Chair
Locations (5):
- United States (5):
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - JHU AVEG, Pittsburgh, Pennsylvania
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington